CLINICAL TRIAL: NCT02271633
Title: The Effect of Nitrate Supplementation: Source of Supplementation
Brief Title: Nitrate Supplementation; Source
Acronym: NO-what
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: METC14-3-020
Record Dates: First submitted 2014-10-13; First posted 2014-10-22 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-05

CONDITIONS: Blood Pressure; Nutritional Physiological Phenomena
Keywords: Nitrate; Bioavailability; Sports
MeSH Terms: interventions — sodium nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sodium nitrate (Active Comparator): Dietary supplement: 800 mg of nitrate in sodium nitrate added with water to get a 140 mL solution (BASF, Ludwigshafen, Germany)
  Interventions: Dietary Supplement: Beetroot juice; Dietary Supplement: Spinach; Dietary Supplement: Rocket salad
- Beetroot juice (Active Comparator): Dietary supplement: 800 mg of nitrate in concentrated beetroot juice (Beet-IT)
  Interventions: Dietary Supplement: Sodium nitrate; Dietary Supplement: Spinach; Dietary Supplement: Rocket salad
- Spinach (Active Comparator): Dietary supplement: 800 mg of nitrate in a spinach based beverage
  Interventions: Dietary Supplement: Sodium nitrate; Dietary Supplement: Beetroot juice; Dietary Supplement: Rocket salad
- Rocket salad (Active Comparator): Dietary supplement: 800 mg of nitrate in a rocket salad based beverage
  Interventions: Dietary Supplement: Sodium nitrate; Dietary Supplement: Beetroot juice; Dietary Supplement: Spinach

INTERVENTIONS:
Dietary Supplement: Sodium nitrate
  Arms: Beetroot juice; Rocket salad; Spinach
Dietary Supplement: Beetroot juice
  Arms: Rocket salad; Sodium nitrate; Spinach
Dietary Supplement: Spinach
  Arms: Beetroot juice; Rocket salad; Sodium nitrate
Dietary Supplement: Rocket salad
  Arms: Beetroot juice; Sodium nitrate; Spinach

SUMMARY:
The main aim of the current study will be to compare the effects of ingesting different nitrate-rich sources on plasma nitrite concentrations.

DETAILED DESCRIPTION:
Oral ingestion of nitrate (NO3-) has been shown to increase plasma nitrate and nitrite levels. Significant lowering of pulmonary oxygen uptake during exercise, as well as significantly lower blood pressure values at rest have been observed after supplementation with nitrate. However, no study has yet described a direct comparison between different nitrate-rich beverages with respect to the bioavailability of nitrate/nitrite and the possible hemodynamic effects. Based on the gaps in current literature, our main goal will therefore be to gain further insight into the effects of nitrate supplementation with different sources on plasma nitrite levels.

ELIGIBILITY:
Inclusion Criteria:

* 18.5 < BMI < 30 kg/m2
* Engagement in regular physical activity ( > 1 h a week)

Exclusion Criteria:

* Use of medication
* Smoking
* Currently supplementing diet with nitrate
* Lactose intolerance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Plasma nitrite levels | Baseline until 5 hours after ingestion
  Plasma nitrite levels following ingestion of dietary nitrate

SECONDARY OUTCOMES:
Plasma levels of nitrate | Baseline until 5 hours post-ingestion
  Plasma nitrate levels following ingestion of dietary nitrate
Resting blood pressure | Baseline, 2.5 hours and 5 hours post-ingestion
  Resting blood pressure measures following ingestion of dietary nitrate
Tongue scraping to assess bacterial mouth flora. | 5 h post-ingestion
  Tongue scraping to assess bacterial mouth flora.

OTHER OUTCOMES:
Baseline characteristics | 1 hour during visit 1 (Screening)
  Resting blood pressure, height, body weight, age, BMI

CONTACTS AND LOCATIONS:
Overall Officials: Lex Verdijk, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Wylie LJ, Kelly J, Bailey SJ, Blackwell JR, Skiba PF, Winyard PG, Jeukendrup AE, Vanhatalo A, Jones AM. Beetroot juice and exercise: pharmacodynamic and dose-response relationships. J Appl Physiol (1985). 2013 Aug 1;115(3):325-36. doi: 10.1152/japplphysiol.00372.2013. Epub 2013 May 2. PMID 23640589
- [Background] van Velzen AG, Sips AJ, Schothorst RC, Lambers AC, Meulenbelt J. The oral bioavailability of nitrate from nitrate-rich vegetables in humans. Toxicol Lett. 2008 Oct 1;181(3):177-81. doi: 10.1016/j.toxlet.2008.07.019. Epub 2008 Aug 3. PMID 18723086
- [Background] Hobbs DA, Kaffa N, George TW, Methven L, Lovegrove JA. Blood pressure-lowering effects of beetroot juice and novel beetroot-enriched bread products in normotensive male subjects. Br J Nutr. 2012 Dec 14;108(11):2066-74. doi: 10.1017/S0007114512000190. Epub 2012 Mar 14. PMID 22414688
- [Background] Liu AH, Bondonno CP, Croft KD, Puddey IB, Woodman RJ, Rich L, Ward NC, Vita JA, Hodgson JM. Effects of a nitrate-rich meal on arterial stiffness and blood pressure in healthy volunteers. Nitric Oxide. 2013 Nov 30;35:123-30. doi: 10.1016/j.niox.2013.10.001. Epub 2013 Oct 10. PMID 24120618
- [Background] Cermak NM, Gibala MJ, van Loon LJ. Nitrate supplementation's improvement of 10-km time-trial performance in trained cyclists. Int J Sport Nutr Exerc Metab. 2012 Feb;22(1):64-71. doi: 10.1123/ijsnem.22.1.64. PMID 22248502
- [Derived] Jonvik KL, Nyakayiru J, Pinckaers PJ, Senden JM, van Loon LJ, Verdijk LB. Nitrate-Rich Vegetables Increase Plasma Nitrate and Nitrite Concentrations and Lower Blood Pressure in Healthy Adults. J Nutr. 2016 May;146(5):986-93. doi: 10.3945/jn.116.229807. Epub 2016 Apr 13. PMID 27075914